CLINICAL TRIAL: NCT02516306
Title: A Phase 1/2 Prospective, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of EV06 Ophthalmic Solution, in Improving Distance Corrected Near Vision in Subjects With Presbyopia
Brief Title: A Study to Evaluate the Safety and Efficacy of EV06 Ophthalmic Solution in Improving Vision in Subjects With Presbyopia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Encore Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EV-C-002
Record Dates: First submitted 2015-07-23; First posted 2015-08-05 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-10

CONDITIONS: Presbyopia
Keywords: Presbyopia; Vision; UNR844
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EV06 Ophthalmic Solution (Experimental): EV06 Ophthalmic Solution: Day 1 - 7 one drop twice per day in one eye; Day 8 - 91 one drop twice per day in both eyes.
  Interventions: Drug: EV06 Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator): Placebo Ophthalmic Solution (EV06 vehicle): Day 1 - 7 one drop twice per day in one eye; Day 8 - 91 one drop twice per day in both eyes.
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: EV06 Ophthalmic Solution
  Other Names: Active treatment
  Arms: EV06 Ophthalmic Solution
Drug: Placebo Ophthalmic Solution
  Other Names: Inactive control (vehicle)
  Arms: Placebo Ophthalmic Solution

SUMMARY:
The purpose of this study is to determine whether EV06 Ophthalmic Solution is safe and effective in improving distance corrected near vision in people who have presbyopia.

DETAILED DESCRIPTION:
Study subjects who were eligible for enrollment and had provided written informed consent were randomized in a 2:1 ratio to use of either EV06 Ophthalmic Solution or Placebo Ophthalmic Solution. For the first 7 days of study product administration (Period 1: Days 1-7), subjects applied 1 drop of their assigned study product to one eye twice per day. For the next 84 days (Period 2: Days 8 - 91), if there were no unanticipated and no significant adverse events observed in the treated eye, subjects applied 1 drop of their assigned study product to both eyes twice per day.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 55 years of age
* Distance Corrected Near Visual Acuity worse than 20/40
* Best Corrected Distance Visual Acuity of 20/20 or better in each eye
* Willing and able to sign consent, following study instructions

Exclusion Criteria:

* Certain pupillary conditions
* Significant astigmatism, glaucoma, diabetes, cataracts, eye surgery, ocular trauma or accommodative issues
* contact lens wear within 3 days prior to and for duration of study
* use of prohibited medications
* participation in a clinical study within 30 days prior

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Expert Clinical Project Lead Ophthalmology, Study Director — Encore Vision, Inc.
Locations (4):
- United States (4):
  - Sall Research Medical Center, Inc., Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Total Eye Care, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- EVO6 Ophthalmic Solution: EV06 Ophthalmic Solution: Day 1 - 7 one drop twice per day in one eye; Day 8 - 91 one drop twice per day in both eyes.
- Placebo: Placebo Ophthalmic Solution: Day 1 - 7 one drop twice per day in one eye. Day 8 - 91 one drop administered twice per day in both eyes.
Period: Period 1: Day 1 - 7
Arm/Group | EVO6 Ophthalmic Solution | Placebo
Started | 50 | 25
Completed | 50 | 25
Not Completed | 0 | 0
Period: Period 2: Day 8 - 91
Arm/Group | EVO6 Ophthalmic Solution | Placebo
Started | 50 | 25
Completed | 49 | 23
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- EV06 Ophthalmic Solution: EV06 Ophthalmic Solution: Period 1 (Day 1 - 7) one drop in one eye twice per day for 7 days; Period 2 (Day 8 - 91) one drop in both eyes twice per day for 84 days.
- Placebo: Placebo Ophthalmic Solution: Period 1 (Day 1 - 7) one drop in one eye twice per day for 7 days; Period 2 (Day 8 - 91) one drop in both eyes twice per day for 84 days.
- Total: Total of all reporting groups
Arm/Group | EV06 Ophthalmic Solution | Placebo | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (3.2) | 51.4 (3.0) | 50.5 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 20 | 53
  Male | 17 | 5 | 22
Region of Enrollment [Number; unit: participants]
  United States | 50 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Ocular Comfort Assessment Following Instillation at Baseline and the Day Prior to Each Study Visit
Description: Ocular comfort was assessed at Baseline (Day 1) and following the last dose on the day prior to each office visit. Comfort was assessed by each subject marking a visual analog scale labeled "0" (Very Comfortable), "5" (Comfortable) and "10" (Very Uncomfortable) immediately following instillation of their assigned study product to one eye (Baseline) or both eyes (Days 8 - 91). A small number indicated better comfort. No formal inferential statistics hypotheses were tested.
Time Frame: Baseline, Day 7, Day 14, Day 30, Day 60, Day 90
Population: Includes all subjects who completed the study: EV06 Ophthalmic Solution (49 of 50) and Placebo Ophthalmic Solution (23 of 25)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EVO6 Ophthalmic Solution: EV06 Ophthalmic Solution: Period 1 (Day 1 - 7) one drop twice per day in one eye; Period 2 (Day 8 - 91) one drop twice per day in both eyes.
- Placebo Ophthalmic Solution: Placebo Ophthalmic Solution: Period 1 (Day 1 - 7) one drop twice per day in one eye; Period 2 (Day 8 - 91) one drop twice per day in both eyes.
Arm/Group | EVO6 Ophthalmic Solution | Placebo Ophthalmic Solution
Number analyzed (Participants) | 49 | 23
units on a scale
  Day 1 | 3.2 (2.4) | 3.3 (2.5)
  Day 7 | 2.4 (2.4) | 2.2 (2.2)
  Day 14 | 2.2 (2.2) | 2.3 (2.2)
  Day 30 | 2.4 (2.0) | 2.2 (2.2)
  Day 60 | 2.1 (2.1) | 3.0 (2.5)
  Day 90 | 2.1 (2.4) | 2.1 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire duration of the study: Day 1 through 91.
Groups:
- EVO6: EV06 Ophthalmic Solution: Period 1 (Day 1 - 7) one drop twice per day to one eye; Period 2 (Day 8 - 91) one drop twice per day to both eyes.
- Placebo: Placebo Ophthalmic Solution: Period 1 (Day 1 - 7) one drop twice per day to one eye; Period 2 (Day 8 - 91) one drop twice per day to both eyes.
Arm/Group | EVO6 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/25
Other Adverse Events (participants affected / at risk) | 18/50 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO6 (N=50) | Placebo (N=25)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Eye irritation (Eye disorders) | 3 (3) | 0 (0)
Instillation site pain (General disorders) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Disgeusia (Nervous system disorders) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less